CLINICAL TRIAL: NCT01722526
Title: An Open-label, Multicenter, Ascending Dose Study of the Tolerability and Safety of Recombinant Human Acid Sphingomyelinase (rhASM) in Patients With Acid Sphingomyelinase Deficiency (ASMD)
Brief Title: Tolerability and Safety Study of Recombinant Human Acid Sphingomyelinase in Acid Sphingomyelinase Deficiency Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI13412; 2012-003542-32 (EudraCT Number); SPHINGO00812 (Other: Genzyme)
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Human Acid Sphingomyelinase Deficiency
Keywords: Human acid sphingomyelinase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant human acid sphingomyelinase (Experimental): Participants will receive rhASM of an initial dose of 0.1 mg/kg, followed by several dose escalations, as tolerated, up to 3.0 mg/kg. All doses are given 2 weeks apart.
  Interventions: Drug: Recombinant human acid sphingomyelinase

INTERVENTIONS:
Drug: Recombinant human acid sphingomyelinase — Administered intravenously every 2 weeks for 26 weeks
  Other Names: GZ402665

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetic, and pharmacodynamic profile of rhASM in adult patients with Acid Sphingomyelinase Deficiency (ASMD) following repeated-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented non-neuronopathic acid sphingomyelinase deficiency
* The patient has a diffusing capacity of carbon monoxide (DLco) >20% and ≤80% of the predicted normal value.
* The patient has a spleen volume ≥6 multiples of normal(MN). A partial splenectomy will be permitted if performed ≥1 year prior to Screening/Baseline and residual spleen volume is ≥6 MN.
* The patient who is receiving lipid lowering therapy should be on a stable dose and regimen of lipid-lowering therapy(ies) for at least 12 weeks prior to Screening/Baseline, with the patient expected to remain on the same dose and regimen throughout the 26-week treatment period.
* The patient who is female and of childbearing potential must have a negative serum pregnancy test for β-HCG.

Exclusion Criteria:

* The patient is female and pregnant or lactating.
* The patient has a Body Mass Index(BMI)>30.
* The patient has received an investigational drug within 30 days prior to study enrollment
* The patient has a medical condition or any extenuating circumstance that may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities.
* The patient has had a major organ transplant
* ALT or AST >250 IU/L or total bilirubin >1.5 mg/dL.
* The patient is unwilling or unable to abstain from the use of alcohol for 1 day prior to and 3 days after each rhASM infusion for the duration of the study.
* The patient requires medications that may decrease rhASM
* The patient is unwilling or unable to avoid the use of medications or herbal supplements that may cause or prolong bleeding, or have potential hepatotoxicity within 10 days prior to and 3 days after liver biopsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Summary of Adverse Events (AEs) | at least 26 weeks

SECONDARY OUTCOMES:
Pharmacokinetics as measured by peak plasma concentration (Cmax), time to peak concentration (tmax), area under curve (AUC), half life (t1/2), drug clearance (CL), and volume of distribution (Vss) | up to 26 weeks
Pharmacodynamics as measured by liver and skin biopsies, plasma, and dried blood spot | up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- Mount Sinai School of Medicine, New York, New York, United States
- St. Mary's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Thurberg BL, Diaz GA, Lachmann RH, Schiano T, Wasserstein MP, Ji AJ, Zaher A, Peterschmitt MJ. Long-term efficacy of olipudase alfa in adults with acid sphingomyelinase deficiency (ASMD): Further clearance of hepatic sphingomyelin is associated with additional improvements in pro- and anti-atherogenic lipid profiles after 42 months of treatment. Mol Genet Metab. 2020 Sep-Oct;131(1-2):245-252. doi: 10.1016/j.ymgme.2020.06.010. Epub 2020 Jun 24. PMID 32620536
- [Derived] Thurberg BL, Wasserstein MP, Jones SA, Schiano TD, Cox GF, Puga AC. Clearance of Hepatic Sphingomyelin by Olipudase Alfa Is Associated With Improvement in Lipid Profiles in Acid Sphingomyelinase Deficiency. Am J Surg Pathol. 2016 Sep;40(9):1232-42. doi: 10.1097/PAS.0000000000000659. PMID 27340749
- [Derived] Wasserstein MP, Jones SA, Soran H, Diaz GA, Lippa N, Thurberg BL, Culm-Merdek K, Shamiyeh E, Inguilizian H, Cox GF, Puga AC. Successful within-patient dose escalation of olipudase alfa in acid sphingomyelinase deficiency. Mol Genet Metab. 2015 Sep-Oct;116(1-2):88-97. doi: 10.1016/j.ymgme.2015.05.013. Epub 2015 May 30. PMID 26049896